CLINICAL TRIAL: NCT02416206
Title: A Phase II Trial of High-dose Bendamustine, Etoposide, Cytarabine, and Melphalan (BeEAM) in the Up-front Treatment of Multiple Myeloma
Brief Title: High Dose Chemotherapy Using BeEAM for Autologous Transplant in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1107
Record Dates: First submitted 2015-03-11; First posted 2015-04-14 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; hematopoietic stem cell transplant
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BeEAM (Experimental): Bendaumustine, Etoposide, Cytrabine and Melphalan in autologous transplant for multiple myeloma
  Interventions: Drug: BeEAM

INTERVENTIONS:
Drug: BeEAM — BeEAM

SUMMARY:
High-dose chemotherapy and autologous stem cell transplantation (ASCT) as part of the up-front treatment of patients with multiple myeloma has been associated with improved disease-free and overall survival in multiple large randomized controlled trials. Following 3-6 cycles of standard induction therapy with biologic agents, consolidation with high dose Melphalan and ASCT has become the standard-of-care approach for fit myeloma patients up to 70 years of age. Single-agent high-dose Melphalan (200mg/m2) is currently the standard-of-care preparative regimen prior to autologous transplant in Myeloma. Historical studies utilizing Busulfan- or Total Body Irradiation-based preparative regimens have yielded similar results to single-agent Melphalan with higher toxicity.

DETAILED DESCRIPTION:
Myeloma patients, following up-front induction therapy, will receive an ASCT following a high-dose bendamustine-based preparative regimen (BeEAM). The primary endpoint of this trial will be the rate of CR at day 100 post-transplant. Experience from the literature, as well as results from our institution, suggests that following ASCT for the upfront treatment of myeloma, the rate of CR at day 100 post-transplant is approximately 45%. It is hoped that under this protocol, this rate will be at least 65%. Thus we statistically formalize this study by testing the null hypothesis that p, the CR rate is 0.65 or more versus the alternative hypothesis that p is less than 0.45. A sample size of 65 pts gives 90% power with an alpha=0.05, using the formula for a one sample binomial (two-sided) test of a proportion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 70 years
* Karnofsky status ≥ 70%
* Diagnosis of Multiple Myeloma
* Within 9 months of the start of induction chemotherapy and no evidence of relapse or progression.
* Availability of Cryopreserved peripheral blood stem cells with a CD34 dose of at least 2x106/kg.

Exclusion Criteria:

* Poor cardiac function: left ventricular ejection fraction <40%
* Poor pulmonary function: FEV1, FVC, or DLCO <40% predicted
* Poor liver function: bilirubin >2.5 mg/dl (not due to hemolysis, Gilbert's or primary malignancy), AST/ALT > 3X ULN
* Poor renal function: Creatinine >2.0 mg/dl or creatinine clearance < 40 mL/min (calculated creatinine clearance is permitted)
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
* Women of childbearing potential who currently are pregnant or who are not practicing adequate contraception
* Patients who have any debilitating medical or psychiatric illness which would preclude their giving informed consent or their receiving optimal treatment and follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Solomon, MD, Principal Investigator — Northside Hospital
Locations (1):
- Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia, United States

REFERENCES:
- [Background] Attal M, Harousseau JL. The role of high-dose therapy with autologous stem cell support in the era of novel agents. Semin Hematol. 2009 Apr;46(2):127-32. doi: 10.1053/j.seminhematol.2009.02.006. PMID 19389496
- [Background] Harousseau JL, Attal M, Divine M, Marit G, Leblond V, Stoppa AM, Bourhis JH, Caillot D, Boasson M, Abgrall JF, et al. Autologous stem cell transplantation after first remission induction treatment in multiple myeloma. A report of the French Registry on Autologous Transplantation in Multiple Myeloma. Stem Cells. 1995 Aug;13 Suppl 2:132-9. doi: 10.1002/stem.5530130721. PMID 8520502
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Harousseau JL, Avet-Loiseau H, Attal M, Charbonnel C, Garban F, Hulin C, Michallet M, Facon T, Garderet L, Marit G, Ketterer N, Lamy T, Voillat L, Guilhot F, Doyen C, Mathiot C, Moreau P. Achievement of at least very good partial response is a simple and robust prognostic factor in patients with multiple myeloma treated with high-dose therapy: long-term analysis of the IFM 99-02 and 99-04 Trials. J Clin Oncol. 2009 Dec 1;27(34):5720-6. doi: 10.1200/JCO.2008.21.1060. Epub 2009 Oct 13. PMID 19826130
- [Background] Kyle RA, Rajkumar SV. Criteria for diagnosis, staging, risk stratification and response assessment of multiple myeloma. Leukemia. 2009 Jan;23(1):3-9. doi: 10.1038/leu.2008.291. Epub 2008 Oct 30. PMID 18971951
- [Background] Alexanian R, Weber D, Giralt S, Dimopoulos M, Delasalle K, Smith T, Champlin R. Impact of complete remission with intensive therapy in patients with responsive multiple myeloma. Bone Marrow Transplant. 2001 May;27(10):1037-43. doi: 10.1038/sj.bmt.1703035. PMID 11438818
- [Background] Alvares CL, Davies FE, Horton C, Patel G, Powles R, Sirohi B, Zuha R, Gatt A, Saso R, Treleaven JG, Dearden CE, Potter MN, Ethell ME, Morgan GJ. Long-term outcomes of previously untreated myeloma patients: responses to induction chemotherapy and high-dose melphalan incorporated within a risk stratification model can help to direct the use of novel treatments. Br J Haematol. 2005 Jun;129(5):607-14. doi: 10.1111/j.1365-2141.2005.05514.x. PMID 15916682
- [Background] Bjorkstrand B, Goldstone AH, Ljungman P, Brandt L, Brunet S, Carlson K, Prentice G, Cavo M, Samson D, de Laurenzi A, et al. Prognostic factors in autologous stem cell transplantation for multiple myeloma: an EBMT Registry Study. European Group for Bone Marrow Transplantation. Leuk Lymphoma. 1994 Oct;15(3-4):265-72. doi: 10.3109/10428199409049723. PMID 7866274
- [Background] Krejci M, Buchler T, Hajek R, Svobodnik A, Krivanova A, Pour L, Adam Z, Mayer J, Vorlicek J. Prognostic factors for survival after autologous transplantation: a single centre experience in 133 multiple myeloma patients. Bone Marrow Transplant. 2005 Jan;35(2):159-64. doi: 10.1038/sj.bmt.1704728. PMID 15543200
- [Background] O'Shea D, Giles C, Terpos E, Perz J, Politou M, Sana V, Naresh K, Lampert I, Samson D, Narat S, Kanfer E, Olavarria E, Apperley JF, Rahemtulla A. Predictive factors for survival in myeloma patients who undergo autologous stem cell transplantation: a single-centre experience in 211 patients. Bone Marrow Transplant. 2006 Apr;37(8):731-7. doi: 10.1038/sj.bmt.1705307. PMID 16501593
- [Background] Giralt S, Vesole DH, Somlo G, Krishnan A, Stadtmauer E, Mccarthy P, Pasquini MC; Blood and Marrow Transplant Clinical Trials Network Multiple Myeloma Working Group. Re: Tandem vs single autologous hematopoietic cell transplantation for the treatment of multiple myeloma: a systematic review and meta-analysis. J Natl Cancer Inst. 2009 Jul 1;101(13):964; author reply 966-7. doi: 10.1093/jnci/djp126. Epub 2009 Jun 17. No abstract available. PMID 19535777
- [Background] Harousseau JL, Moreau P. Evolving role of stem cell transplantation in multiple myeloma. Clin Lymphoma Myeloma. 2005 Sep;6(2):89-95. doi: 10.3816/CLM.2005.n.034. PMID 16231846
- [Background] Lahuerta JJ, Grande C, Martinez-Lopez J, De La Serna J, Toscano R, Ortiz MC, Larregla S, Conde E, Insunza A, Gonzalez-San Miguel JD, Bargay J, Cabrera R, Garcia-Ruiz JC, Albo C, Garcia-Alonso L, Solano F, Vivancos P, Leon A, San Miguel J; Grupo Espanol de Sindromes Linfoproliferativos/Trasplante Autologo de Medula Osea. Tandem transplants with different high-dose regimens improve the complete remission rates in multiple myeloma. Results of a Grupo Espanol de Sindromes Linfoproliferativos/Trasplante Autologo de Medula Osea phase II trial. Br J Haematol. 2003 Jan;120(2):296-303. doi: 10.1046/j.1365-2141.2003.04067.x. PMID 12542490
- [Background] Anagnostopoulos A, Aleman A, Ayers G, Donato M, Champlin R, Weber D, Alexanian R, Giralt S. Comparison of high-dose melphalan with a more intensive regimen of thiotepa, busulfan, and cyclophosphamide for patients with multiple myeloma. Cancer. 2004 Jun 15;100(12):2607-12. doi: 10.1002/cncr.20294. PMID 15197803
- [Background] Brinker BT, Waller EK, Leong T, Heffner LT Jr, Redei I, Langston AA, Lonial S. Maintenance therapy with thalidomide improves overall survival after autologous hematopoietic progenitor cell transplantation for multiple myeloma. Cancer. 2006 May 15;106(10):2171-80. doi: 10.1002/cncr.21852. PMID 16598756
- [Background] Desikan KR, Tricot G, Dhodapkar M, Fassas A, Siegel D, Vesole DH, Jagannath S, Singhal S, Mehta J, Spoon D, Anaissie E, Barlogie B, Munshi N. Melphalan plus total body irradiation (MEL-TBI) or cyclophosphamide (MEL-CY) as a conditioning regimen with second autotransplant in responding patients with myeloma is inferior compared to historical controls receiving tandem transplants with melphalan alone. Bone Marrow Transplant. 2000 Mar;25(5):483-7. doi: 10.1038/sj.bmt.1702167. PMID 10713623
- [Background] Shimoni A, Smith TL, Aleman A, Weber D, Dimopoulos M, Anderlini P, Andersson B, Claxton D, Ueno NT, Khouri I, Donato M, Korbling M, Alexanian R, Champlin R, Giralt S. Thiotepa, busulfan, cyclophosphamide (TBC) and autologous hematopoietic transplantation: an intensive regimen for the treatment of multiple myeloma. Bone Marrow Transplant. 2001 Apr;27(8):821-8. doi: 10.1038/sj.bmt.1703007. PMID 11477439
- [Background] Christoforidou AV, Saliba RM, Williams P, Qazilbash M, Roden L, Aleman A, Weber D, Mendoza F, Podoloff D, Wendt R 3rd, Breitz H, Alexanian R, Champlin R, Giralt S. Results of a retrospective single institution analysis of targeted skeletal radiotherapy with (166)Holmium-DOTMP as conditioning regimen for autologous stem cell transplant for patients with multiple myeloma. Impact on transplant outcomes. Biol Blood Marrow Transplant. 2007 May;13(5):543-9. doi: 10.1016/j.bbmt.2006.12.448. Epub 2007 Feb 26. PMID 17448913
- [Background] Giralt S, Bensinger W, Goodman M, Podoloff D, Eary J, Wendt R, Alexanian R, Weber D, Maloney D, Holmberg L, Rajandran J, Breitz H, Ghalie R, Champlin R. 166Ho-DOTMP plus melphalan followed by peripheral blood stem cell transplantation in patients with multiple myeloma: results of two phase 1/2 trials. Blood. 2003 Oct 1;102(7):2684-91. doi: 10.1182/blood-2002-10-3250. Epub 2003 May 1. PMID 12730103
- [Background] Moreau P, Facon T, Attal M, Hulin C, Michallet M, Maloisel F, Sotto JJ, Guilhot F, Marit G, Doyen C, Jaubert J, Fuzibet JG, Francois S, Benboubker L, Monconduit M, Voillat L, Macro M, Berthou C, Dorvaux V, Pignon B, Rio B, Matthes T, Casassus P, Caillot D, Najman N, Grosbois B, Bataille R, Harousseau JL; Intergroupe Francophone du Myelome. Comparison of 200 mg/m(2) melphalan and 8 Gy total body irradiation plus 140 mg/m(2) melphalan as conditioning regimens for peripheral blood stem cell transplantation in patients with newly diagnosed multiple myeloma: final analysis of the Intergroupe Francophone du Myelome 9502 randomized trial. Blood. 2002 Feb 1;99(3):731-5. doi: 10.1182/blood.v99.3.731. PMID 11806971
- [Background] Grey-Davies E, Bosworth JL, Boyd KD, Ebdon C, Saso R, Chitnavis D, Mercieca JE, Morgan GJ, Davies FE. Bendamustine, Thalidomide and Dexamethasone is an effective salvage regimen for advanced stage multiple myeloma. Br J Haematol. 2012 Feb;156(4):552-5; author reply 555. doi: 10.1111/j.1365-2141.2011.08887.x. Epub 2011 Sep 26. No abstract available. PMID 21950692
- [Background] Lentzsch S, O'Sullivan A, Kennedy RC, Abbas M, Dai L, Pregja SL, Burt S, Boyiadzis M, Roodman GD, Mapara MY, Agha M, Waas J, Shuai Y, Normolle D, Zonder JA. Combination of bendamustine, lenalidomide, and dexamethasone (BLD) in patients with relapsed or refractory multiple myeloma is feasible and highly effective: results of phase 1/2 open-label, dose escalation study. Blood. 2012 May 17;119(20):4608-13. doi: 10.1182/blood-2011-12-395715. Epub 2012 Mar 26. PMID 22451423
- [Background] Ludwig H, Kasparu H, Leitgeb C, Rauch E, Linkesch W, Zojer N, Greil R, Seebacher A, Pour L, Weissmann A, Adam Z. Bendamustine-bortezomib-dexamethasone is an active and well-tolerated regimen in patients with relapsed or refractory multiple myeloma. Blood. 2014 Feb 13;123(7):985-91. doi: 10.1182/blood-2013-08-521468. Epub 2013 Nov 13. PMID 24227817
- [Background] Ponisch W, Heyn S, Beck J, Wagner I, Mohren M, Hoffmann FA, Lange T, Schmalfeld M, Zehrfeld T, Schwarzer A, Winkelmann C, Edelmann T, Rohrborn R, Hebenstreit K, Al-Ali HK, Jakel N, Niederwieser D. Lenalidomide, bendamustine and prednisolone exhibits a favourable safety and efficacy profile in relapsed or refractory multiple myeloma: final results of a phase 1 clinical trial OSHO - #077. Br J Haematol. 2013 Jul;162(2):202-9. doi: 10.1111/bjh.12361. Epub 2013 May 21. PMID 23692564
- [Background] Ponisch W, Mitrou PS, Merkle K, Herold M, Assmann M, Wilhelm G, Dachselt K, Richter P, Schirmer V, Schulze A, Subert R, Harksel B, Grobe N, Stelzer E, Schulze M, Bittrich A, Freund M, Pasold R, Friedrich T, Helbig W, Niederwieser D; East German Study Group of Hematology and Oncology (OSHO). Treatment of bendamustine and prednisone in patients with newly diagnosed multiple myeloma results in superior complete response rate, prolonged time to treatment failure and improved quality of life compared to treatment with melphalan and prednisone--a randomized phase III study of the East German Study Group of Hematology and Oncology (OSHO). J Cancer Res Clin Oncol. 2006 Apr;132(4):205-12. doi: 10.1007/s00432-005-0074-4. Epub 2006 Jan 10. PMID 16402269
- [Background] Visani G, Malerba L, Stefani PM, Capria S, Galieni P, Gaudio F, Specchia G, Meloni G, Gherlinzoni F, Giardini C, Falcioni S, Cuberli F, Gobbi M, Sarina B, Santoro A, Ferrara F, Rocchi M, Ocio EM, Caballero MD, Isidori A. BeEAM (bendamustine, etoposide, cytarabine, melphalan) before autologous stem cell transplantation is safe and effective for resistant/relapsed lymphoma patients. Blood. 2011 Sep 22;118(12):3419-25. doi: 10.1182/blood-2011-04-351924. Epub 2011 Aug 3. PMID 21816830

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BeEAM
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BeEAM
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 59 [40 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 33
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: To Estimate the Response at Day 100 Following Transplant (Rate of CR)
Description: Using IMWG criteria: PR (partial response) noted as >50% reduction of serum M-protein and reduction in 24hr urinary M-protein by >90% or to <200mg/24h; VgPR (very good partial response) noted as serum and urine M-protein detectable by immunofixation but not on electrophoresis or >90% reduction in serum M-protein plus urine M-protein level <100mg/24h; CR (complete response) noted as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow; sCR (stringent complete response) noted as CR defined above plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | BeEAM
Number analyzed (Participants) | 65
Participants
  Complete Response (CR1) | 26
  Very Good Partial Response (VGPR1) | 32
  Partial Response (PR1) | 7

2. Secondary Outcome: Number of Patients With Overall Survival Post-transplant
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | BeEAM
Number analyzed (Participants) | 65
Participants | 60

3. Secondary Outcome: Number of Patients With Progression-free Survival
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | BeEAM
Number analyzed (Participants) | 65
Participants | 37

4. Secondary Outcome: Number of Patients Who Relapsed After Transplant
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | BeEAM
Number analyzed (Participants) | 65
Participants | 28

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 3 years. Adverse events were assessed up to 3 months
Arm/Group | BeEAM
All-Cause Mortality (participants affected / at risk) | 5/65
Serious Adverse Events (participants affected / at risk) | 48/65
Other Adverse Events (participants affected / at risk) | 17/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeEAM (N=65)
neutropenic fever (Investigations) | 31
Esophagitis (Gastrointestinal disorders) | 17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BeEAM (N=65)
peripheral neuropathy (Nervous system disorders) | 3
hypertension (Cardiac disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT02416206/Prot_SAP_000.pdf